CLINICAL TRIAL: NCT06660394
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Investigate the Efficacy, Safety, and Tolerability of LP352 in the Treatment of Seizures in Children and Adults With Dravet Syndrome
Brief Title: A Phase 3, Placebo-Controlled Study to Investigate LP352 in Children and Adults With Dravet Syndrome (DS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Longboard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP352-302; 2024-514937-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dravet Syndrome
Keywords: Antiseizure medication; Epilepsy; Neurodevelopmental disorders; Developmental and epileptic encephalopathy; LP352; Seizures; DEEp SEA; Bexicaserin
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy; Neurodevelopmental Disorders; Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LP352 (Experimental): Participants will be titrated up to highest tolerated dose of LP352 during the Titration period (Visit 2 - Visit 5), followed by maintenance period (Visit 5 - Visit 8) and then taper/down titration period.
  Interventions: Drug: LP352
- Placebo (Placebo Comparator): Placebo for LP352
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LP352 — LP352 will be administered orally or through G-tube/ percutaneous endoscopic gastrostomy (PEG) tube
  Other Names: Bexicaserin
  Arms: LP352
Drug: Placebo — Participants will be administered with matching placebo orally or through G-tube/ PEG tube
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
This (DEEp SEA Study) is a double-blind, randomized, placebo-controlled, multicenter study to investigate the efficacy, safety, and tolerability of LP352 in the treatment of seizures in children and adults with DS. The study consists of 3 main phases: Screening, Titration period, and Maintenance period, followed by a Taper period and Follow-Up. Participants will be randomized to LP352 or placebo. The total duration of the study will be approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DS must fulfill all of the following criteria:

  1. Participants with seizure onset age >1 and <20 months
  2. The participant has a history of at least 1 of the following seizure type(s): prolonged generalized tonic-clonic, hemiclonic, myoclonic, tonic, atonic, atypical absence, focal impaired awareness, nonconvulsive status epilepticus
* The participant has a current occurrence of at least 1 of the following countable motor seizure types: generalized tonic-clonic, tonic (bilateral), clonic (bilateral), atonic (bilateral) with truncal/leg involvement, focal motor (including hemiclonic), and focal to bilateral tonic-clonic
* The participant has demonstrated an average of at least 4 countable motor seizures per month for the 3 months prior to Screening.
* The participant has been taking 1 to 4 antiseizure medications (ASMs) at a stable dose for at least 4 weeks prior to Screening.
* The participant, parent, or caregiver is willing and able (in the judgment of the investigator) to comply with completion of the diaries throughout the study.
* The participant must be willing and able to provide written informed consent.

Exclusion Criteria:

* The participant has a history of infantile/epileptic spasms.
* The participant has been admitted to a medical facility for treatment of status epilepticus requiring mechanical ventilation within 3 months prior to Screening.
* The participant has a neurodegenerative disorder as indicated by magnetic resonance imaging or genetic testing.
* The participant has an acquired lesion/injury unrelated to the primary etiology that could contribute as a secondary cause of seizures.
* The participant is receiving exclusionary medications.
* The participant has used any cannabis product or cannabidiol that is not in oral solution/capsule/tablet form, not obtained from a government-approved dispensary, or contains ≥50% Delta-9-tetrahydrocannabinol (THC).
* The participant has unstable, clinically significant neurologic (other than the disease being studied, eg, recurrent strokes), psychiatric, cardiovascular (eg, pulmonary arterial hypertension, cardiac valvulopathy, orthostatic hypotension/tachycardia), pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
* The participant is unwilling to comply with any of the study requirements or timelines.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Frequency Percent Change in Countable Motor Seizures During Treatment Compared to Baseline | Baseline and up to 15 Weeks
  The percent change from Baseline in countable motor seizure frequency during Treatment will be calculated as countable motor seizure frequency during Treatment minus countable motor seizure frequency during Screening and divided by seizure frequency during Screening and multiplied by 100 where each seizure frequency will be based on number of seizures.

SECONDARY OUTCOMES:
Safety and Tolerability of LP352 | Up to 21 Weeks
  Safety and tolerability as measured by incidence and severity of non-serious Treatment Emergent Adverse Events (TEAEs), Serious Adverse events (SAEs), AEs leading to discontinuation and clinically significant changes in laboratory parameters (hematology, serum chemistry and Urinalysis), physical examination findings, vital signs, growth parameters (height and weight), 12-lead electrocardiograms (ECGs), C-SSRS responses, and PHQ-9 total score and Question 9 score.
Percentage of participants with ≥ 50% Reduction in countable motor seizures during Treatment compared to Baseline | Baseline and up to 15 Weeks
Frequency Percent Change in Countable Motor Seizures during Maintenance compared to Baseline | Baseline and up to 15 Weeks

CONTACTS AND LOCATIONS:
Locations (77):
- United States (22):
  - Arkansas Children's Hospital - PIN, Little Rock, Arkansas
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - The Stanford Division of Child Neurology, Palo Alto, California
  - UCSF Children's Hospital, San Francisco, California
  - Children's Hospital Colorado., Aurora, Colorado
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Nicklaus Children's Hospital - PIN, Miami, Florida
  - Research Institute of Orlando LLC, Orlando, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Rare Disease Research, LLC - Atlanta - RDR - PIN, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago - PIN, Chicago, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Institute of Neurology and Neurosurgery at Saint Barnabas, LLC, Livingston, New Jersey
  - Northeast Regional Epilepsy Group - Morristown - 310 Madison Ave, Morristown, New Jersey
  - NYU Comprehensive Epilepsy Center - BRANY - PPDS, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Le Bonheur Childrens Outpatient Center - PIN, Memphis, Tennessee
  - Child Neurology Consultants of Austin - 6811 Austin Center Blvd, Austin, Texas
  - Cook Children's Jane and John Justin Neurosciences Center - PIN, Fort Worth, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Multicare Health System - Mary Bridge Pediatrics, Tacoma, Washington
- Australia (8):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - The Alfred Hospital, Melbourne
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - UZ Antwerpen, Antwerp
- Brazil (2):
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto Hospital de Base - PPDS, São José do Rio Preto, São Paulo
  - Instituto de Psiquiatria HC FMUSP, São Paulo
- London Health Sciences Centre -800 Commissioners Rd E, London, Ontario, Canada
- China (4):
  - Peking University First Hospital - Daxing Campus, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Children's Hospital, Capital Medical University - PIN, Beijing
- France (8):
  - Hôpital Roger Salengro, Lille, Nord
  - Hospices Civils de Lyon - Hôpital Pierre Wertheimer, Bron
  - AP-HM- Hôpital de La Timone, Marseille
  - Hôpital Necker - Enfants Malades, Paris
  - AP-HP - Hôpital universitaire Robert-Debré, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (4):
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Gesellschaft für Epilepsieforschung e.V., Bielefeld
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Epilepsie-Zentrum Bodensee, Ravensburg
- Italy (5):
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome, Lazio
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genova
- Japan (3):
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
  - Osaka City General Hospital, Osaka-Shi Miyakojima-Ku, Ôsaka
- Children's Clinical University Hospital, Riga, Latvia
- Portugal (3):
  - ULS de Coimbra, EPE - Hospital Pediátrico de Coimbra, Coimbra
  - ULS de Santa Maria,EPE - Hospital de Santa Maria - PPDS, Lisbon
  - ULS de Santo António, EPE - Centro Materno Infantil Norte, Porto
- Serbia (4):
  - University Clinical Center of Serbia - Dr Subotica 6 - PPDS, Belgrade, Belgrade
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Spain (8):
  - Hospital Sant Joan de Deu - PIN, Espluges de Llobregat, Barcelona
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Málaga
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vithas Madrid La Milagrosa, Madrid
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid
  - Hospital Vithas Malaga, Málaga
- United Kingdom (2):
  - Royal Victoria Infirmary, Newcastle upon Tyne, Northamptonshire
  - Queen Elizabeth University Hospital - PPDS, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided